CLINICAL TRIAL: NCT06295263
Title: Application of AI Technology for the Diagnosis and Treatment of Geriatric Diseases
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202203-028-1
Record Dates: First submitted 2024-02-17; First posted 2024-03-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Alzheimer Disease; Nervous System Diseases; Geriatric Diseases
Keywords: Parkinson Disease; Alzheimer Disease; Nervous System Diseases; geriatric diseases; AI; Deep learning
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Nervous System Diseases | interventions — Gait; Eye Movements; Blood Specimen Collection; Urination; Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — lood, urine, stool, saliva, etc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Parkinson Disease group: 100 patients with primary Parkinson's disease were included, mainly from outpatient clinics and wards of the Parkinson's Disease and Movement Disorders Center. Inclusion criteria: patients with primary Parkinson's disease, based on the 2015 MDS Parkinson's disease diagnostic criteria. Exclusion criteria: ① patients suffering from other central nervous system diseases, such as cerebrovascular disease, traumatic brain injury, central system inflammatory diseases, intracranial tumors and postoperative neurosurgery; ② patients with various types of cognitive disorders (MMSE score <24); ③ severe psychiatric disorders that are difficult to cooperate.
  Interventions: Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers
- Alzheimer Disease group: One hundred patients with Alzheimer's disease were included, mainly from geriatric neurology outpatient clinics and wards (F5A & F6A). Inclusion criteria: patients with Alzheimer's disease, meeting the IWG-2 clinical diagnostic criteria as the basis. Exclusion criteria: ① patients suffering from other central nervous system diseases, such as cerebrovascular disease, traumatic brain injury, central system inflammatory diseases, intracranial tumors and postoperative neurosurgery; ② severe psychiatric illnesses that are difficult to cooperate with.
  Interventions: Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers
- Nervous System Diseases group: Neurodegenerative diseases (non-PD non-AD) group 100: source neurology outpatient clinic visits, exclusion criteria: ① patients suffering from other central nervous system diseases, such as cerebrovascular disease, traumatic brain injury, central system inflammatory diseases, intracranial tumors and neurosurgery postoperative; ② severe psychiatric diseases difficult to cooperate with the person.
  Interventions: Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers
- Healthy geriatric group: Healthy elderly control 80 people, from peer attendees and health checkup centers. Inclusion criteria: ① Voluntary participation in this study and signing of informed consent; ② Age and gender matched with the patients in the case group; Exclusion criteria: ① Previous history of chronic diseases related to the study subjects, such as cerebrovascular disease, traumatic brain injury, inflammatory diseases of the central system, intracranial tumors and neurosurgery, etc.; ② Patients with various types of cognitive disorders (MMSE scores <24); ③ Those with poor adherence.
  Interventions: Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers
- Healthy Adults Group: Young healthy controls 80 people, from peer attendees and health screening centers. Inclusion criteria: ① Voluntary participation in the study and signing of informed consent; ② Gender matched with the patients in the case group, age <60 years; Exclusion criteria: ① History of chronic diseases related to the study subjects, such as cerebrovascular disease, traumatic brain injury, inflammatory diseases of the central system, intracranial tumors and neurosurgery, etc.; ② With various types of cognitive disorders (MMSE scores <24); ③ Poor adherence to the study. Poor adherence.
  Interventions: Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers

INTERVENTIONS:
Other: Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers — Handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers in all experimental and control groups

SUMMARY:
1) Characteristics of handwriting, gait, speech, eye movements, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers in patients with Alzheimer's disease.

(2) Characteristics of handwriting, gait, language, eye movement, biological samples (blood, urine, stool, saliva, etc.), imaging, EEG, and other relevant markers in patients with Parkinson's disease.

(3) Characteristics of handwriting, gait, language, eye movement, biological samples (blood, urine, stool, saliva, etc.), images, EEG, and other relevant markers in patients with other neurological disorders.

(4) Characteristics of handwriting, gait, language, eye movement, biological samples (blood, urine, stool, saliva, etc.), images, EEG and other relevant markers in elderly patients.

DETAILED DESCRIPTION:
1. Study variables (factors) and measurements

1. All enrolled subjects collected data including general clinical information, PD patients completed motor function assessment and non-motor function assessment, AD patients completed cognitive function assessment and mood-sleep assessment, patients with other neurological disorders perfected disease-related clinical information and scale assessment, and healthy elderly and young controls perfected general clinical information and scale screening.
2. All selected subjects complete handwriting recording, gait assessment, language entry and eye movement recording, and collect biological samples (blood (3 ml/case), urine (3 ml/case), stool (2 g/case), saliva (3 ml/case) and other clinical test results), imaging, EEG and other relevant markers for the study of diagnostic and treatment plan and correlation analysis of AI technology.

   1. Motor symptom assessment: UPDRS score
   2. Non-motor symptom assessment: Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MOCA), Hamilton Anxiety Scale (HAMD), and Hamilton Anxiety Diagnostic Scale (HAD). Hamilton Anxiety Scale (HAMD), Hamilton Depression Scale (HDMD), SF-36.

      2. Sample size 100 patients with primary Parkinson's disease were included, 100 patients with Alzheimer's disease were included, 100 patients with other neurological disorders were included, 80 healthy elderly controls, and 80 healthy young controls.

      3 Data collection and management Data collection was firstly collected by applying the paper version of the case report form, and then entered into the computer by a specialized person.

      4. Statistical analysis methods For continuous variables, statistical descriptions were performed using mean ± standard deviation, and for categorical variables, frequency and rate (%) were used. For comparison of parameters between two groups, t-test or rank sum test was used for continuous type variables and chi-square test was used for categorical variables. For one-way correlation analysis, Pearson or Spearman correlation analysis was used. For multifactor analysis, generalized linear model or logistic regression model was used. All of the above parameters were considered statistically significant at p<0.05.

      5. Quality control
      1. Clinical data disease diagnosis: determined by two Parkinson's and movement disorders group deputy chief physicians and above;
      2. Scale assessment: adjudicated by two scale-trained neurologists;
      3. Statistics: performed by clinical statisticians. 6. Research feasibility analysis Qilu Hospital of Shandong University is a one-stop diagnosis and treatment center for Parkinson's disease and a clinical research center of geriatrics in Shandong Province, with a large patient attendance group and clear clinical significance; our research center is equipped with handwriting analyzer, gait analyzer, speech and eye movement capture analyzer, and has analyzers for collecting biological samples, imaging information and EEG information, which has the basis for further in-depth research.

ELIGIBILITY:
1. Inclusion Criteria 1.1 A total of 100 patients with primary Parkinson's disease were enrolled. The inclusion criteria were as follows: patients with primary Parkinson's disease, based on the 2015 MDS diagnostic criteria for Parkinson's disease. Disorder (MMSE score < 24); (3) those with severe mental illness who are difficult to cooperate.

   1.2 A total of 100 patients with Alzheimer's disease were enrolled. The inclusion criteria were as follows: patients with Alzheimer's disease, based on the IWG-2 clinical diagnostic criteria.

   1.3 Neurodegenerative diseases (non-PD and non-AD) group (n = 100) : meeting the diagnostic criteria of the corresponding diseases.

   1.4 Eighty healthy elderly controls were included. The inclusion criteria were as follows: ① voluntarily participated in this study and signed the informed consent; ② Age and gender were matched with the case group.

   1.5 80 young healthy controls, inclusion criteria: ① voluntarily participated in this study and signed the informed consent; ② Gender was matched with the case group, and the age was less than 60 years old.
2. Exclusion Criteria 2.1 A total of 100 patients with PD were enrolled. Exclusion criteria: ① patients with other central nervous system diseases, such as cerebrovascular diseases, brain trauma, inflammatory diseases of the central system, intracranial tumors and after neurosurgery; ② patients with various types of cognitive impairment (MMSE score < 24); (3) those with severe mental illness who are difficult to cooperate.

2.2 A total of 100 patients with Alzheimer's disease were enrolled. The exclusion criteria were: ① patients with other central nervous system diseases, such as cerebrovascular diseases, brain trauma, central system inflammatory diseases, intracranial tumors and after neurosurgery; ② patients with severe mental illness who are difficult to cooperate.

2.3 Neurodegenerative diseases (non-PD non-AD) group (n = 100), exclusion criteria: ① patients with other central nervous system diseases, such as cerebrovascular diseases, brain trauma, central system inflammatory diseases, intracranial tumors and after neurosurgery; ② patients with severe mental illness who are difficult to cooperate.

2.4 Eighty healthy elderly controls were included. The exclusion criteria were as follows: ① History of chronic diseases related to the study subjects, such as cerebrovascular diseases, brain trauma, inflammatory diseases of the central system, intracranial tumors and neurosurgery; ② patients with various types of cognitive impairment (MMSE score < 24); ③ Poor compliance.

2.5 80 young healthy controls, exclusion criteria: ① history of chronic diseases related to the study subjects, such as cerebrovascular diseases, brain trauma, inflammatory diseases of the central system, intracranial tumors and neurosurgical surgery; ② patients with various types of cognitive impairment (MMSE score < 24); ③ Poor compliance.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. 100 patients with primary Parkinson's disease were included, mainly from the outpatient clinics and wards of the Parkinson's Disease and Movement Disorders Center. Inclusion criteria: patients with primary Parkinson's disease, based on the 2015 MDS Parkinson's disease diagnostic criteria.
  2. 100 patients with Alzheimer's disease were included, mainly from geriatric neurology outpatient clinics and wards (F5A&F6A). Inclusion criteria: patients with Alzheimer's disease, meeting the IWG-2 clinical diagnostic criteria as the basis.
  3. Neurodegenerative diseases (non-PD and non-AD) group 100 people: the source of neurology outpatient clinic
  4. 80 healthy elderly controls, from peer attendees and health check centers.
  5. 80 young healthy controls, from peer clinic attendees and health screening centers.
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Handwriting | 2022-2~2026-6
  The patterns and related auxiliary features of patients' handwritten notes were analyzed,the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.
gait | 2022-2~2026-6
  The patients' stride length and gait frequency were analyzed，the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.
speech | 2022-2~2026-6
  The speech of the patients were collected and analyzed,the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.
eye movements | 2022-2~2026-6
  The eye movement data of the patients were collected and analyzed,the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.
biological samples (blood, urine, stool, saliva, etc.) | 2022-2~2026-6
  3-5ml of biological specimens were retained for testing and data analysis
images | 2022-2~2026-6
  MRI、MRA、SWI、DTI and other imaging data were analyzed,the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.
EEG | 2022-2~2026-6
  Mean frequency, relative power, absolute power, electrode correlation, coherence, time-frequency analysis，etc
other relevant markers | 2022-2~2026-6
  Some other markers are waiting to be studied and discovered,the specific indicators used should be adjusted according to the results of artificial intelligence calculation, and the unit should be adjusted according to the indicators used.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No